CLINICAL TRIAL: NCT01409278
Title: The Evaluation of the Efficacy of Local Infiltration Analgesia and Infusion for Total Hip Arthroplasty
Brief Title: Local Anesthetic Infiltration and Infusion for Pain Control After Hip Replacement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Trinity Health Of New England (Other)
Responsible Party: Sanjay Sinha, Saint Francis Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 09-07-002
Record Dates: First submitted 2011-08-02; First posted 2011-08-04 (Estimated); Last update posted 2011-08-04 (Estimated); Status verified 2009-08

CONDITIONS: Osteoarthritis
MeSH Terms: conditions — Osteoarthritis | interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Ropivacaine infiltration and infusion. (Experimental): Ropivicaine infiltration followed by continuous ropivicaine infusion for 48 hours.
  Interventions: Procedure: Ropivacaine infiltration and infusion.
- Ropivacaine and Saline (Experimental): Ropivicaine infiltration followed by normal saline infusion.
  Interventions: Procedure: Ropivacaine infiltration and saline infusion.
- Saline infiltration and infusion. (Placebo Comparator): Normal saline infiltration followed by saline infusion.
  Interventions: Procedure: Normal Saline

INTERVENTIONS:
Procedure: Ropivacaine infiltration and saline infusion. — 50ml ropivacaine 0.2% with keterolac 15mg infiltration followed by normal saline infusion at 5ml per hour
  Arms: Ropivacaine and Saline
Procedure: Ropivacaine infiltration and infusion. — 50 ml infiltration of ropivacaine 0.2% and ketorolac 15mg admixture followed by ropivacaine 0.2 % at 5ml per hour infusion for 48 hours.
  Arms: Ropivacaine infiltration and infusion.
Procedure: Normal Saline — 50ml of normal saline infiltration followed by normal saline infusion at 5ml per hour
  Arms: Saline infiltration and infusion.

SUMMARY:
The purpose of this study is to examine three different ways to control pain after hip replacement:

1. One time injection of ropivacaine before wound closure
2. One time injection of ropivacaine before wound closure plus slow release of ropivacaine via catheter for 48 hours
3. Standard practice of patient controlled pump

ELIGIBILITY:
Inclusion Criteria:

* total knee replacement

Exclusion Criteria:

* History of neurological disease, diabetes, pregnancy, allergy to local anesthetic solutions chronic narcotic use ability to consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2009-08; Primary Completion 2010-07 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
The pain medication requirement for 48 hours after surgery in three groups. | 48 hours after surgery

SECONDARY OUTCOMES:
Pain scores, incidence of nausea and vomiting and patient satisfaction in each group. | 48 hours after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Sanjay Sinha, M.D., Principal Investigator — Saint Francis Hospital
Locations (1):
- Saint Francis Hospital and Medical Center, Hartford, Connecticut, United States